CLINICAL TRIAL: NCT05865535
Title: A Phase 1B Dose Escalation Study of AV-380 in Combination With Standard of Care Chemotherapy in Metastatic Cancer Patients With Cachexia and Elevated GDF-15 Levels
Brief Title: A Dose Escalation Study of AV-380 in Cancer Patients With Cachexia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AV-380-22-102
Record Dates: First submitted 2023-05-02; First posted 2023-05-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Cohorts (Experimental): Experimental: Dose escalation cohorts of AV-380 administered by IV infusion
  Interventions: Biological: AV-380

INTERVENTIONS:
Biological: AV-380 — AV-380 is an immunoglobulin (Ig) G1 monoclonal antibody (mAb) intended to bind circulating human growth differentiation factor 15 (GDF-15), a cytokine involved in cancer-induced cachexia.

SUMMARY:
This open label ascending dose study is designed to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of AV-380 in cancer patients with Cachexia. AV-380 is an immunoglobulin (Ig) G1 monoclonal antibody (mAb) intended to bind circulating human growth differentiation factor 15 (GDF-15), a cytokine involved in cancer-induced cachexia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years of age at the time of signing the informed consent.
2. Patients with histologically confirmed solid tumor cancer who are actively receiving SoC therapy for this cancer.
3. Patients with cachexia as defined by Fearon criteria:

   1. Weight loss > 5% over past 6 months (in absence of simple starvation), or
   2. BMI < 20 kg/m2 and any degree of weight loss > 2%, or
   3. Sarcopenia and any degree of weight loss > 2%
4. Patients with life expectancy ≥ 3 months

Exclusion Criteria:

1. History of allergic or anaphylactic reaction to any monoclonal antibody (IgG protein) or molecules made of components of monoclonal antibody
2. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 2 weeks before first dose of study treatment.
3. Myocardial infarction or heart failure of New York Heart Association Grade 3-4 within 3 months prior to start of protocol therapy
4. Uncontrolled pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
5. Cachexia is caused by other reasons (e.g., severe chronic obstructive pulmonary disease, heart failure, or HIV/AIDS), or the patient has uncontrolled reversible causes of reduced oral food intake, including, but not limited to, oral mucositis, nausea/vomiting, diarrhea, and/or obstruction, impairing the patient's ability to eat as determined by the Investigator.
6. Patients receiving tube feedings or parenteral nutrition at the time of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) | From enrollment to the last follow-up visit approximately 60-days post dose
  AEs as characterized by incidence, type, frequency, and severity (graded according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE])
Toxicity | While receiving study drug (up to 4 months)
  Dose-limiting Toxicity (DLT) events observed at increasing doses of AV-380
Laboratory Abnormalities | From enrollment to the last follow-up visit approximately 60-days post dose.
  Laboratory abnormalities as characterized by type, frequency, severity (graded according to NCI-CTCAE v5.0) and timing.

SECONDARY OUTCOMES:
Cmax | From first dose to the last follow-up visit approximately 60-days post dose.
  Maximum observed plasma concentration for AV-380
Tmax | From first dose to the last follow-up visit approximately 60-days post dose
  Time to reach the Cmax for AV-380
AUC(0-t) | From first dose to the last follow-up visit approximately 60-days post dose.
  Area under the plasma concentration-time curve from zero time to the last measurable point for AV-380

OTHER OUTCOMES:
Immunogenicity | From first dose to the last follow-up visit approximately 60-days post dose.
  Serum levels of Anti-Drug Antibody (ADA) against AV-380 and their potential relationship with AEs and serum levels of GDF-15
Weight | From enrollment to the last follow-up visit approximately 60-days post dose.
  Change from baseline body weight during the study
Patient-Reported Outcomes | From enrollment to the end of treatment, approximately 4 months
  Change from baseline in the following questionnaires: Functional Assessment of Anorexia Cachexia Therapy (FAACT); Patient global impression of severity (PGI-S) and patient global impression of change (PGI-C) for appetite, fatigue, and physical activity.
Lumbar (L3) Skeletal Muscle Index (L3SMI) | From enrollment to the end of treatment, approximately 4 months
  Measurement of a cross-sectional area of muscle at the level of the third lumbar vertebra (L3) using computed tomography (CT) scan
Physical Function | From enrollment to the end of treatment, approximately 4 months
  Change from baseline in physical function endpoints, including Short Physical Performance Battery test and digital measures of non-sedentary time
Serum level of GDF-15 | From enrollment to the last follow-up visit approximately 60-days post dose.
Albumin and CRP | From enrollment to the last follow-up visit approximately 60-days post dose.
  Change from baseline in albumin and CRP levels
Tumor status | From enrollment to the last follow-up visit approximately 60-days post dose.
  Evaluate the effect of AV-380 on tumor burden and tumor status, per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1)
Biomarkers | From first dose to the last follow-up visit approximately 60-days post dose.
  including activin A and cytokine levels (e.g., monocyte chemoattractant protein-1 [MCP-1] and proinflammatory)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Cancer and Blood Specialty Clinic, Lakewood, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Hartford Hospital, Hartford, Connecticut
  - Advent Health Orlando Hospital, Orlando, Florida
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - New York Cancer And Blood Specialists, Shirley, New York
  - Oregon Health and Science University, Portland, Oregon
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Community Clinical Trials, Kingwood, Texas

IPD SHARING:
Plan to Share IPD: No